CLINICAL TRIAL: NCT00869479
Title: Validation of a Questionnaire as a Screening Tool to Identify Signs and Symptoms of Nephrogenic Systemic Fibrosis
Brief Title: Validation of a Questionnaire to Identify Signs and Symptoms of Nephrogenic Systemic Fibrosis
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Alexandra Kimball, MD, Massachusetts General Hospital
Other Study IDs: 2008P002371
Record Dates: First submitted 2009-03-17; First posted 2009-03-26 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Nephrogenic Systemic Fibrosis
Keywords: Nephrogenic Systemic Fibrosis; Screening
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: subjects with a histologically-proven diagnosis of NSF
- 2: subjects with other fibrosing skin diseases
- 3: subjects with non-fibrosing skin diseases
- 4: subjects without skin diseases

SUMMARY:
The Primary Aim of this study is to validate a questionnaire as a screening tool to identify subjects with symptoms suggestive of nephrogenic systemic fibrosis (NSF). The investigators believe that there will be difference between subjects with NSF and other skin conditions and normal skin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age or older.
2. Willing and able to understand and provide oral informed consent.
3. Able to complete study and comply with study procedures.

Exclusion Criteria:

1. Subject is unable to provide oral consent.
2. Psychiatric or other conditions which might, in the opinion of the Principal Investigator, interfere with study evaluations or pose a risk to subject safety during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Massachusetts General Hospital Dermatology and Rheumatology clinics
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Difference in the number of "yes" answers between NSF subjects and subjects with non-fibrosing skin diseases or without skin diseases. | 1 day

SECONDARY OUTCOMES:
Similarity in answers between NSF subjects and subjects with other fibrosing skin diseases. | 1 day
Sensitivity of the questionnaire when applied to NSF subjects. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kay, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Todd DJ, Kay J. Nephrogenic systemic fibrosis: an epidemic of gadolinium toxicity. Curr Rheumatol Rep. 2008 Jul;10(3):195-204. doi: 10.1007/s11926-008-0033-6. PMID 18638427
- [Background] Todd DJ, Kagan A, Chibnik LB, Kay J. Cutaneous changes of nephrogenic systemic fibrosis: predictor of early mortality and association with gadolinium exposure. Arthritis Rheum. 2007 Oct;56(10):3433-41. doi: 10.1002/art.22925. PMID 17907148
- [Derived] Lima XT, Alora-Palli MB, Kimball AB, Kay J. Validation of a screening instrument for nephrogenic systemic fibrosis. Arthritis Care Res (Hoboken). 2013 Apr;65(4):637-42. doi: 10.1002/acr.21877. PMID 23097320